CLINICAL TRIAL: NCT04972760
Title: Baricitinib in Patients With Relapsing or naïve Dermatomyositis: a Multicenter Randomized Controlled Trial (BIRD)
Brief Title: Baricitinib in Patients With Relapsing or naïve Dermatomyositis
Acronym: BIRD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP180612; 2020-004987-24 (EudraCT Number)
Record Dates: First submitted 2021-06-14; First posted 2021-07-22 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Dermatomyositis
Keywords: Dermatomyositis; baricitinib; steroid sparing
MeSH Terms: conditions — Dermatomyositis | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- baricitinib arm (Experimental): Patients receive baricitinib plus prednisone taper plus one immunosuppressive drug (either methotrexate or azathioprine) for a duration of 24 weeks. Corticosteroids are tapered following a predefined protocol.
  Interventions: Drug: Baricitinib
- placebo arm (Placebo Comparator): Patients receive placebo plus prednisone taper plus one immunosuppressive drug (either methotrexate or azathioprine) for a duration of 24 weeks. Corticosteroids are tapered following a predefined protocol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Baricitinib, 4 mg/d, oral route for 24 weeks
  Arms: baricitinib arm
Drug: Placebo — Placebo, 4 mg/d, oral route for 24 weeks
  Arms: placebo arm

SUMMARY:
Dermatomyositis (DM) is a rare and disabling condition with an important impairment of quality of life and possible life-threatening complications.

Treatment is based on high doses of corticosteroids but this exposes patients to adverse events (cardiovascular mortality, glucocorticoids-induced muscle and skin damages). Corticosteroids taper is associated with disease relapses. Although there is no evidence from the literature, clinical practice guidelines recommends the use of DMARDs such as methotrexate. However, response is not complete and these DMARDS take time to act.

The interferon type I (IFN-I) pathway is involved in the pathophysiology of DM. Janus kinase 1 and 2 transduces IFN-I signals. In addition, JAK2 inhibition enhances muscle repair and force generation.

JAK 1/2 inhibitors permitted to dramatically and rapidly improve relapsing DM patients (n=4, case series).

Our hypothesis is that Janus kinase 1 and 2 (JAK1/2) inhibitors (baricitinib) will permit to obtain dermatomyositis (DM) improvement with a steroid sparing effect as compared to usual care.

Our primary objective is to evaluate the efficacy of baricitinib (JAK1/2 inhibitor) to obtain prednisone-free moderate improvement (ACR/EULAR ≥ 40) of DM as compared to placebo in addition to usual care.

BIRD is a multicenter phase III double blind randomized placebo-controlled trial with two parallel arms (1:1). This is an add-on trial to usual care with rapid corticoid taper.

This is a multicenter trial in different medical departments in hospitals across France in different regions.

Out- and in patients will be recruited in hospital departments involved in management and diagnosis of DM: departments of dermatology, rheumatology and internal medicine.

DETAILED DESCRIPTION:
Dermatomyositis (DM) is a rare and disabling condition with an important impairment of quality of life and possible life-threatening complications.

Treatment is based on high doses of corticosteroids but this exposes patients to adverse events (cardiovascular mortality, glucocorticoids-induced muscle and skin damages). Corticosteroids taper is associated with disease relapses. Although there is no evidence from the literature, clinical practice guidelines recommends the use of DMARDs such as methotrexate. However, response is not complete and these DMARDS take time to act.The interferon type I (IFN-I) pathway is involved in the pathophysiology of DM. Janus kinase 1 and 2 transduces IFN-I signals. In addition, JAK2 inhibition enhances muscle repair and force generation .

JAK 1/2 inhibitors permitted to dramatically and rapidly improve relapsing DM patients (n=4, case series) .

BIRD is a multicenter phase III double blind randomized placebo-controlled trial with two parallel arms (1:1). This is an add-on trial to usual care with rapid corticoid taper. Both groups (experimental and control groups) will receive corticosteroids and the conventional immunosuppressive drug (either azathioprine or methotrexate)

Our primary objective is to evaluate the efficacy of baricitinib (JAK1/2 inhibitor) to obtain prednisone-free DM moderate improvement as compared to placebo, in addition to usual care.

Primary endpoint: moderate improvement (defined as a total improvement score superior or equal to 40 following ACR/EULAR definition) without corticosteroids at week 24 (prednisone-free moderate improvement).

This multicenter trial involves different medical departments in hospitals across France in different regions. Out- and in patients will be recruited in hospital departments involved in management and diagnosis of DM: departments of dermatology, rheumatology and internal medicine.

Eligible patients will sign a written informed consent after full oral and written information about the trial. They will be randomized in 1:1 ratio to receive baricitinib plus prednisone taper plus one immunosuppressive drug (either methotrexate or azathioprine) (experimental group) or placebo plus prednisone taper plus one immunosuppressive drug (either methotrexate or azathioprine) (control group) for a duration of 24 weeks. In both groups, corticosteroids are tapered following a predefined protocol.

5 visits are planned:

* screening visit (W-4 to D-1)
* baseline visit (W0)
* follow-up visit 1 (W5 +/-5 days)
* follow-up visit 2 (W12 +/-5 days)
* end of study visit 3 (W24+/-5 days) Data will be collected by investigator and clinical research associate on an electronic case report form (eCRF) via a web browser.

The primary analysis will be the comparison between experimental and control groups of the rate of prednisone-free moderate improvement at 24 weeks in the intent to treat population. In order to demonstrate a difference in the rate of primary outcome at 24 weeks from 30% in the control group to 70% in the experimental group, with a power of 80%, a bilateral alpha risk of 5%, and a 15% rate of loss of follow-up, 62 patients are necessary.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥ 18 years old) < 65 years old
* Dermatomyositis defined according to the 239th ENMC criteria either naïve or non-naïve DM
* Active disease (ACR/EULAR criteria) defined as :

  * Manual Muscle Testing (MMT-8) <145/150 and at least two additional abnormal corset measurements (CSM): >3/10 cm on Visual Analogue Scale (VAS) of patient global, physician global and extra-muscular disease activity, Health Assessment Questionnaire Disability Index >0.25, or elevated muscle enzymes.
  * Or cutaneous CDASI > 20 and at least two additional abnormal corset measurements (CSM): >3/10 cm on Visual Analogue Scale (VAS) of patient global, physician global and extra-muscular disease activity, Health Assessment Questionnaire Disability Index >0.25, or elevated muscle enzymes
* for relapsing/non naïve DM patients :

  * in case of corticosteroid exposure patient must receive a stable dose < 30 mg/d prednisone with or without additional immunosuppressive therapy for at least 4 weeks before the baseline visit.
  * Stable dose of immunosuppressive therapy for at least 3 months before
* Affiliation to a social security regime
* Written informed consent

Exclusion Criteria:

* Life-threatening complications :

  * Severe swallowing troubles defined as: food swallowed the wrong way and/or time to drink a glass of 200 ml water above 30 seconds related to DM.
  * Interstitial lung disease related to the DM with one among the following complications (complications must be related to the ILD): dyspnea NYHA III, hypoxemia with PaO2≤65 mmHg, and/or DLCOc/Alveolar Volume ≤70% (pulmonary function test)
  * Symptomatic myocarditis o Loss of walking ability
* Patient with deep vein thrombosis/pulmonary embolism or antecedent
* Patient with antecedent of cardiovascular event (myocardial infarction or ischemic stroke)
* Patient who is current or past long-time smoker
* Pregnant or lactating, or women planning to become pregnant or initiating breastfeeding
* No effective contraception during the study and one week after for women of childbearing age
* Renal impairment defined as clearance < 60 ml
* Strong Organic Anion Transporter 3 (OAT3) inhibitors
* Active cancer or history of malignancy
* Active severe infection including active hepatitis
* Evidence of latent tuberculosis (as documented by a positive QuantiFERON-TB Gold plus test)
* Absolute Neutrophil Count < 1x109 cells/L
* Haemoglobin (Hb) < 8 g/dL
* Severe hepatic impairment attested by FV (coagulation factor)<30%
* Liver insufficiency (Prothrombin time <60%)
* Previous treatment exposure defined as follow : • Rituximab treatment within 6months before inclusion

  * IVIg, or cyclophosphamide infusion within the month before inclusion
  * both methotrexate (0.3 mg/kg/w) and azathioprine exposure for at least 3 months each and at the 0.3 mg/kg/w and 2-3 mg/kg/d dosages respectively with failure of both (but exposure and/or failure to either of these two drugs alone is not an exclusion criterion)
  * for naïve DM patients only, more than 2 weeks treatment duration with corticosteroids at the dose of 1 mg/kg/d before the inclusion.
* Hypersensitivity to the active substance (baricitinib) or to any of the excipients
* Contraindication to Methotrexate and/or Azathioprine including hypersensitivity to the active substances or to any of the excipients
* Conditions affecting the outcomes (Expected poor compliance)
* Severe disease damages: e.g. muscle weakness mainly related to muscle damage such as fat replacement of muscle) defined as persistent changes in anatomy, physiology, pathology or function which result from previously active disease and from complications of therapy or other events (e.g.; muscle atrophy, fatty replacement; skin scars, poikiloderma ). Severe disease damage is considered when the patient condition has no or minor ability to improve with the treatment.
* Significant uncontrolled cardiovascular, cerebrovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neuropsychiatric disorders, or abnormal laboratory values that developed during a qualifying study that, in the opinion of the investigator, poses an unacceptable risk for the patient's participation
* Chest imaging (CT scan or radiograph) showing abnormalities not related with the DM in the last 12 weeks judged by the investigator as clinically significant.
* Participants included in other intervention research involving humans
* Patient under tutorship or guardianship, and incapable to give informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Moderate improvement at 24 weeks without prednisone: prednisone-free moderate improvement. | 24 weeks
  The rate of patients with a moderate improvement at 24 weeks, defined as a total improvement score superior or equal to 40 following ACR/EULAR definition. The investigator will consider that patients following the planned prednisone tapering scheme (corticosteroids 0 mg/d at W24) will be prednisone-free.

SECONDARY OUTCOMES:
Dermatomyositis minimal improvement | 5, 12 and 24 weeks
  The rate of patients with a minimal improvement, defined as a total improvement score ≥20 points (ACR/EULAR definition)
Dermatomyositis moderate improvement | 5, 12 and 24 weeks
  The rate of patients with a moderate improvement, defined as a total improvement score ≥40 points (ACR/EULAR definition)
Dermatomyositis major improvement | 5, 12 and 24 weeks
  The rate of patients with a major improvement, defined as a total improvement score ≥60 points (ACR/EULAR definition)
Primary endpoint prednisone-free moderate improvement at Weeks 24 in subgroups | 24 weeks
  * DM naive patients at baseline vs others
  * DM with a severe muscle weakness (MMT8 baseline <125/150) vs others
Cutaneous disease activity and damage | 5, 12 and 24 weeks
  Cutaneous disease activity and damage evaluated using the Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) - Activity and CDASI damages (from 0 to 48, 48 is the maximum disease severity)
Cumulative incidence of relapse | up to 24 weeks
  Cumulative incidence of relapse with the time to first relapse
Cumulative dose of corticosteroids | 24 weeks
  Cumulative dose of corticosteroids at 24 weeks
Average prednisone dose per day through the last 4 weeks (0 mg per day, of more than 0 mg to not more than 4.0 mg per day, of more than 4.0 mg to not more than 7.5 mg per day, and of more than 7.5 mg per day). | 24 weeks
  Proportion of participants with an average prednisone dose of 0 mg per day, of more than 0 mg to not more than 4.0 mg per day, of more than 4.0 mg to not more than 7.5 mg per day, and of more than 7.5 mg per day through the last 4 weeks.
Adverse events | up to 24 weeks
  Incidence, nature, and severity of adverse events and serious adverse events and laboratory abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: YVES ALLENBACH, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitie-Salpêtrière hospital APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodological sound proposal.